CLINICAL TRIAL: NCT00144846
Title: A Randomized, Double-Blind, Parallel-group, Multi-Center Study of Albuterol Sulfate HFA Inhalation Aerosol Delivered Cumulatively With a Valved Holding Chamber and an Attached Facemask in Subjects Between Birth to 23 Months of Age With Acute Wheezing Due to Obstructive Airways Disease
Brief Title: Inhaled Albuterol Sulfate For Acute Wheezing Due To Obstructive Airways Disease In Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB030002
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: wheezing; bronchospasm; albuterol sulfate HFA
MeSH Terms: conditions — Asthma; Respiratory Sounds; Bronchial Spasm

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: albuterol sulfate inhalation aerosol

INTERVENTIONS:
Drug: albuterol sulfate inhalation aerosol

SUMMARY:
This study evaluates the effect of cumulative dose administration of albuterol sulfate inhalation aerosol delivered with valved holding chamber and facemask. This is a four week study in birth to 23 month old subjects who are experiencing acute wheezing due to obstructive airways disease.

ELIGIBILITY:
Inclusion criteria:

* Must be an outpatient.
* Age at second visit must be birth to <24 months old.
* Parent/guardian who is willing to sign, or has signed, an informed consent.
* Must have acute wheezing consistent with reversible obstructive airway disease.
* Must have an asthma symptoms score between 4-9 based on the TAL score (Modified Tal Asthma Symptoms Score measured by the study site) at Screening (Visit 1) while the subject is breathing room air.

Exclusion criteria:

* History of life-threatening asthma or wheezing that requires admission to an intensive care unit for treatment within 3 months prior to Screening, or he/she has been treated in the emergency room and admitted to the hospital for airways obstruction on two or more occasions within 3 months prior to Screening, or there is a history of intubation for respiratory distress due to airways obstruction.
* Has impending respiratory failure.
* Taken medications such as acute/chronic systemic corticosteroids, CNS stimulants, investigational medications, theophylline or aminophylline, anti-arrhythmic within a certain time period prior to the study.
* Having the following signs or symptoms: 1)present with fever (rectal temperature >100.5 ºF or tympanic temperature >101.5ºF); 2) present with known pulmonary (lung) and/or cardiac (heart) congenital malformations; 3) have an underlying chronic disease (respiratory (Chronic pulmonary disease includes congenital anomalies, bronchopulmonary dysplasia, and cystic fibrosis), cardiac, renal, or liver insufficiency, immunodeficiency, encephalopathy); 4) known or suspected foreign body aspiration; 5) their Modified Tal Asthma Symptoms Score is 10; 6) their weight is below a certain limit for the average for their age; 8) they were born before 34 weeks' gestation. 9) Laboratory tests for serum potassium and blood glucose within the following limits (potassium between 3.0-5.8 mEq/L and glucose between 45-140mg/dL).

Max Age: 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2004-09; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To evaluate safety (adverse events, vital signs, physical exams, ECG monitoring etc.) of cumulative dosing of albuterol sulfate inhalation aerosol

SECONDARY OUTCOMES:
To assess the efficacy measures (percent change from baseline over entire treatment period in the TAL score, respiratory rate, wheezing etc.) of cumulative dosing of albuterol sulfate inhalation aerosol.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (29):
- United States (27):
  - GSK Investigational Site, Hoover, Alabama
  - GSK Investigational Site, Fort Mohave, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Alhambra, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, DeKalb, Illinois
  - GSK Investigational Site, Mandeville, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Alliance, Nebraska
  - GSK Investigational Site, Johnson City, New York
  - GSK Investigational Site, Utica, New York
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Huber Heights, Ohio
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Vienna, Virginia
- Puerto Rico (2):
  - GSK Investigational Site, Hato Rey, Puerto Rico
  - GSK Investigational Site, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Abstract submitted to AAAAI 2007: Efficacy of Ventolin( HFA MDI cumulative dosing in children <24 months old. AM Davis, MD, W Lincourt, BS, R Trivedi, MS, A Ellsworth, BS, C Crim, MD. GlaxoSmithKline, RTP, NC
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: SB030002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SB030002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SB030002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SB030002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SB030002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SB030002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SB030002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register